CLINICAL TRIAL: NCT04183608
Title: An Open-label Randomized Trial COmparing staNdard of Care Versus Treat to Target With telemonitoRing and Patient Education in Patients With Ulcerative cOlitis Initiating adaLimumab: The CONTROL Trial
Brief Title: A Trial COmparing staNdard of Care Versus Treat to Target With telemonitoRing and Patient Education in Patients With Ulcerative cOlitis Initiating Adalimumab
Acronym: CONTROL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GETAID-2018-01
Record Dates: First submitted 2019-10-28; First posted 2019-12-03 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Ulcerative Colitis
Keywords: IBD; UC
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Standard of care (Active Comparator): In standard of care, patient only visits every 3 months the doctor so the optimization of treatment can be done only at this frequency.
  Interventions: Drug: Adalimumab
- Groupe T2T with telemonitoring and patient education (Active Comparator): Treatment with e-Monitoring, home fecal calprotectin testing and therapy education.
  Interventions: Drug: Adalimumab; Diagnostic Test: Calprotectin; Other: e-Monitoring; Other: Therapy Education

INTERVENTIONS:
Drug: Adalimumab — Patients will all receive Adalimumab 160/80/40mg EOW until V1 (W14) followed by 40mg EOW until V2 (W26)
Diagnostic Test: Calprotectin — Fecal calprotectin dosing at home with IBDoc
  Arms: Groupe T2T with telemonitoring and patient education
Other: e-Monitoring — e-Monitoring at Week 6, Week 10, Week 14, Week 18, Week 22, Week 26, Week 34, Week 38, Week 42 and Week 48
  The patient must complete the first 2 questions of the Mayo score:
  * Stool frequency
  * The frequency of bleeding
  He must also complete the information on his injections
  Arms: Groupe T2T with telemonitoring and patient education
Other: Therapy Education — Patient Education at W0, W2, W14, W26 and W38.
  Arms: Groupe T2T with telemonitoring and patient education

SUMMARY:
PHASE: IV

DESCRIPTIVE: Randomized, interventional, open label multicenter trial

POPULATION: Moderate to severe ulcerative colitis

STUDY TREATMENTS: Patients will all receive Adalimumab 160/80/40mg EOW until V1 (W14) followed by 40mg EOW until V2 (W26) and could be optimized up to 80mg EOW (or 40 EW according to patient and/or investigator preference) for two months and then could be optimized up to 80mg EOW (or 40 EW according to patient and/or investigator preference) and azathioprine (2.0/2.5 mg/kg/ day) or methotrexate (25 mg EW) until V3 (W 38).

OBJECTIVES: To assess the impact of a treat to target treatment follow up by e-Monitoring and fecal calprotectin dosing at home associated to an appropriate patient education versus standard treatment follow up at W48 in patients requiring a treatment with adalimumab (Humira®).

DETAILED DESCRIPTION:
NUMBER OF PATIENTS : 238 patients in 20 sites in France

RECRUITMENT PERIOD : The trial duration for each patient will be 144 weeks

MAIN ENDPOINT : At week 48 success defined by: Endoscopic remission defined by an endoscopic Mayo score 0

SECONDARY ENDPOINTS:

At W48

* Clinical remission (Clinical remission is defined as a total Mayo score ≤2 points, with no individual sub score >1, and a Mayo endoscopy sub score of 0 or 1)
* Remission without steroids
* Endoscopic healing rate with Mayo score 0 or 1
* UCEIS score
* Histological healing (Nancy score)
* Remission rate and remission rate without steroids at study visits and W48
* Quality of life evolution (evaluate visit W0 vs W14, W26, W38 and W48)
* Patients satisfaction
* Continuous response
* Safety and tolerability
* Anti-TNF pharmacokinetics
* Number of visits in trial
* Number of UC related hospitalizations
* Number of colectomies
* Treatment compliance (questionnaire)
* Patient adhesion (questionnaire)
* Medico-economic analysis

ELIGIBILITY:
Inclusion Criteria:

* Adults with moderately-to-severely active Ulcerative Colitis (UC) who had an inadequate response to or failed to tolerate steroids and thiopurines (azathioprine or 6-mercaptopurine), methotrexate or vedolizumab or adults with moderately-to-severely active UC who had no response to an adequate steroid course
* Age ≥ 18 years and < 75 years
* Patients scheduled to start a treatment with adalimumab
* Naïve to anti-TNF therapy and other biologics known to be effective for UC (approved or investigational) except for vedolizumab
* Naïve to JAK inhibitors (approved or investigational)
* Moderately-to-severely active UC for at least 3 months with a Mayo score of 6-12 points (endoscopy subscore of at least 2)
* Established diagnosis of UC for at least 3 months (pancolitis, left-sided colitis, proctosigmoiditis and proctitis are allowed).
* Patient has to be treated with oral 5-ASA at time of inclusion regardless of the dose if no contra-indication.
* Azathioprine, 6-mercaptopurine or methotrexate will be stopped two weeks before inclusion.
* A contraceptive method during the whole trial for childbearing potential female
* Patient familiar with Smartphone and internet use

Exclusion Criteria:

* Patients unable to give their consent (because of their physical or mental state).
* Absence of written consent.
* Pregnancy or breastfeeding.
* Patients with severe acute colitis or patients at imminent risk for colectomy.
* History of colectomy.
* History of colonic mucosal dysplasia or adenomatous colonic polyps that are not removed.
* Screening stool trial positive for enteric pathogens or Clostridium difficile toxin.
* Oral corticosteroids at a dose > 40 mg prednisone or its equivalent per day at inclusion (oral steroids should be at stable dose at least 7 days before inclusion)
* Any current or previous use of cyclosporine, tacrolimus, anti-TNF therapy, and other biologics (except vedolizumab), JAK inhibitors (approved or investigational), or any current or previous use of an investigational agent within 5 half-lives of that agent before the first trial agent injection.
* Contraindication to anti-TNF therapy according to drug labeling:

  * Active infection.
  * Non-treated latent tuberculosis.
  * Heart failure (NYHA: Grade III and IV).
  * Malignancy during the previous 5 years.
  * Demyelinating neurological disease.
  * Current or recent (less than 4 weeks) vaccination with attenuated live vaccines
* Patients with a dominant arm deficiency or physical impairment impeding the achievement of the tests
* Patients using a prohibited medication
* Patients participating in another trial or being in a follow-up period for another trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2020-01-14 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Endoscopic Remission | Week 48
  Treatment success of a treat to target with telemonitoring follow up using e-Monitoring and fecal calprotectin dosing at home associated to an appropriate patient education compared to standard treatment follow up at Week 48.
  Definition of treatment success: Endoscopic remission defined by an endoscopic Mayo score 0

SECONDARY OUTCOMES:
Efficacy of adalimumab treatment on clinical remission (at Week 48) | Week 48
  * Remission without steroids:
  * Remission rate and remission rate without steroids at study visits and Week 48
Efficacy of adalimumab treatment on endoscopic Healing (at Week 48) | Week 48
  Endoscopic healing rate with Mayo score 0 or 1
Efficacy of adalimumab treatment on endoscopic mucosal healing | Week 48
  UCEIS score
Efficacy of adalimumab treatment on histological Healing (at Week 48) | Week 48
  Histological healing (Nancy index)
Efficacy of adalimumab treatment on patient quality of life (at Week 48) | Week 48
  Quality of life evolution (evaluate visit 0 vs -Week 14, Week 26, Week 38 and Week 48)
Patient satisfaction | Week 48
  Patient satisfaction evaluate with all questionnaires of quality of life
Treatment compliance | Week 48
  Treatment compliance evaluate at every visit
Patient adhesion | Week 48
  Patient adhesion evaluate with questionnaire
Disability score evolution | Week 48
  IBD Disability index, evaluate visit 0 vs - Week 14, Week 26, Week 38 and Week 48
Medico-economic analysis | Week 48
  Medico-economic comparative analysis between standard of care follow up and tight monitoring follow up
Continuous Clinical Response (CCR) | Week 48
  Definition: Partial Mayo Response at each visit (Visit 1, Visit 2, Visit 3) with a total Mayo response on Week 48 Visit 4 visit. In the telemonitoring group the partial Mayo limited to questions 1 and 2 will be directly answered by patients themselves through ePRO2 they will score the first 2 questions of partial Mayo from home and send that info to the investigator.
Loss of clinical response | Week 48
  Pharmacokinetic dosage of Adalimumab (Anti-TNF)
Number of visits in trial | Week 48
  Number of visits in trial per patients
Colectomies at Week 48 | Week 48
  Proportion of patients with colectomy
UC related Hospitalizations at Week 48 | Week 48
  Proportion of UC related hospitalizations

CONTACTS AND LOCATIONS:
Locations (24):
- France (24):
  - Centre hospitalier de Cholet, Cholet, Maine Et Loire
  - CHU Amiens- Picardie (site Sud), Amiens
  - CHRU de Besançon - Hôpital Jean Minjoz, Besançon
  - CHU Caen Hôpital Côte de Nacre, Caen
  - CHU Estaing, Clermont-Ferrand
  - APHP - Hôpital Beaujon, Clichy
  - CH Colmar - Hôpital Pasteur, Colmar
  - Centre hospitalier de Douai, Douai
  - CHRU Lille Hôpital Claude Huriez, Lille
  - APHM - Hôpital Nord, Marseille
  - GHI Le Raincy-Montfermeil, Montfermeil
  - CHU Montpellier - Hôpital Saint Eloi, Montpellier
  - CHU Nantes - Hôpital Hotel Dieu, Nantes
  - CHU Nice- Hopital l'Archet, Nice
  - CHU Nîmes - Hôpital Universitaire Caremeau, Nîmes
  - CHU Bordeaux - Hôpital Haut Lévêque, Pessac
  - CHU Lyon Sud, Pierre-Bénite
  - CHU Rennes Hôpital Pontchaillou, Rennes
  - CH Saint Etienne Hopital Nord, Saint-Priest-en-Jarez
  - CH Toulon - CHITS CH Sainte Musse, Toulon
  - CHU Toulouse - Hôpital Rangueil, Toulouse
  - CH Tourcoing - Hôpital Gustave Dron, Tourcoing
  - CHU Nancy - Hôpital de Brabois, Vandœuvre-lès-Nancy
  - APHP - Hôpital du Kremlin-Bicêtre, Le Kremlin-Bicêtre, Île-de-France Region

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391